CLINICAL TRIAL: NCT04319172
Title: Multicentric Study of Coronavirus Disease 2019 (COVID-2019) in Solid Organ Transplant Recipients
Acronym: COVIDSOT
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Network for Research in Infectious Diseases (Other); Grupo de Estudio de la Infección en el Trasplante (GESITRA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVIDSOT
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Transplant Recipient; Infections, Coronavirus
Keywords: Transplant Recipient; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Biochemical analysis
  * Hemogram
  * Microbiological testing will be made: blood culture, pleural liquid culture, gram stain and culture of sputum, detection of pneumococcus and Legionella pneumophila antigen in urine, in cases of pneumonia.
  * Nasopharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall purpose of this project is to better understand the incidence, risk factors, etiology, clinical manifestations and outcome of tCOVID19 in solid organ transplant recipients. The results obtained will allow us to gain insight on the need of antiviral treatment, on the strategy for complications surveillance, on how to adjust the immunosuppressant therapy and on the level of care in which each patient should be treated. In order to attain the objectives previously described we will develop a multicenter prospective study of consecutive cases of COVID-19 among solid organ transplant recipients.

DETAILED DESCRIPTION:
There will be a clinical follow-up of the patients included in this study to observe possible complications and survival rate. Data collected form this study will be evaluated with a descriptive statistical analysis of the cohort consisting of analysis of the risk factors of COVID-19. Subsequently a multivaried logistic regression analysis will be performed in which the factors selected from the analysis and those clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 16 years with a solid organ transplant diagnosed of COVID-19.

NOTE: A confirmed case of infection, is defined by a clinical syndrome that is compatible to that of an respiratory infection (fever, cough and/or dyspnea) and the presence of a positive microbiological result.

Exclusion Criteria:

* Absence of informed consent after giving the information regarding the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 16 years with a solid organ transplant diagnosed of COVID-19.
Sampling Method: Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of coronavirus infection in Solid Organ Transplant Recipients | From baseline at the time of signature of informed consent form to day 28 after confirmation of positive test to coronavirus
  Number of Solid Organ Transplant Recipients positive to coronavirus
Clinical manifestations of coronavirus infection in Solid Organ Transplant Recipients | From baseline at the time of signature of informed consent form to day 28 after confirmation of positive test to coronavirus
  Number of participants who present clinical symptoms possibly related to coronavirus infection in Solid Organ Transplant Recipients
Presence of other risk factors | From baseline at the time of signature of informed consent form to day 28 after confirmation of positive test to coronavirus
  Gathering possible risk factors in coronavirus infection in Solid Organ Transplant
Establish the frequency and type of complications related to the net state of the patient immunosuppression | From baseline at the time of signature of informed consent form to day 28 after confirmation of positive test to coronavirus
  Establish the frequency and type of complications related to the net state of the patient immunosuppression

SECONDARY OUTCOMES:
Frequency of co-infections | From baseline at the time of signature of informed consent form to day 28 after confirmation of positive test to coronavirus
  Another infections at the time of coronavirus positive infection will be gathered
Mortality | From baseline at the time of signature of informed consent form up to study completion at 3 months folllow-up
  Number of deaths caused or complicated by coronavirus infection in patients who has recceived Solid Organ Transplant
Laboratory characteristics | At inclusion and at 28 days of follow up
  Biochemical analysis, hemogram,
Determination of coronavirus viral load | At inclusion at 14 days and at 28 days
  Nasopharyngeal swabs
Microbiological testing | At inclusion at 14 days and at 28 days
  According to the clinical manifestations at blood culture, pleural liquid culture, gram stain and culture of sputum, detection of pneumococcus and Legionella pneumophila antigen in urine, in cases of pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Cordero-Matía, MD-PhD, Study Chair — University Hospital Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Planning for the study will be shared with potential sites pertaining to Spanish Network for Research in Infectious Disease (REIPI) and Group for the Study of Infection in Transplantation and the Immunocompromised Host (GESITRA-IC) for participation. IPD is not foreseen out of this groups due to the specific characteristics of patients and sites to be candidates for study participation.
Supporting Information: Study Protocol, ICF
Time Frame: One year after the initiation of the study
Access Criteria: Spanish Network for Research in Infectious Disease (REIPI) and Group for the Study of Infection in Transplantation and the Immunocompromised Host (GESITRA-IC)

REFERENCES:
- [Background] Cordero E, Perez-Romero P, Moreno A, Len O, Montejo M, Vidal E, Martin-Davila P, Farinas MC, Fernandez-Sabe N, Giannella M, Pachon J; Novel influenza A(H1N1) Study Group of Spanish Network for Research in Infectious Diseases (REIPI). Pandemic influenza A(H1N1) virus infection in solid organ transplant recipients: impact of viral and non-viral co-infection. Clin Microbiol Infect. 2012 Jan;18(1):67-73. doi: 10.1111/j.1469-0691.2011.03537.x. Epub 2011 Jul 25. PMID 21790857
- [Background] Peghin M, Los-Arcos I, Hirsch HH, Codina G, Monforte V, Bravo C, Berastegui C, Jauregui A, Romero L, Cabral E, Ferrer R, Sacanell J, Roman A, Len O, Gavalda J. Community-acquired Respiratory Viruses Are a Risk Factor for Chronic Lung Allograft Dysfunction. Clin Infect Dis. 2019 Sep 13;69(7):1192-1197. doi: 10.1093/cid/ciy1047. PMID 30561555
- [Background] Eichenberger EM, Soave R, Zappetti D, Small CB, Shore T, van Besien K, Douglass C, Westblade LF, Satlin MJ. Incidence, significance, and persistence of human coronavirus infection in hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2019 Jul;54(7):1058-1066. doi: 10.1038/s41409-018-0386-z. Epub 2018 Nov 1. PMID 30385869
- [Background] Pinana JL, Madrid S, Perez A, Hernandez-Boluda JC, Gimenez E, Terol MJ, Calabuig M, Navarro D, Solano C. Epidemiologic and Clinical Characteristics of Coronavirus and Bocavirus Respiratory Infections after Allogeneic Stem Cell Transplantation: A Prospective Single-Center Study. Biol Blood Marrow Transplant. 2018 Mar;24(3):563-570. doi: 10.1016/j.bbmt.2017.11.001. Epub 2017 Nov 15. PMID 29155041
- [Background] Garbino J, Crespo S, Aubert JD, Rochat T, Ninet B, Deffernez C, Wunderli W, Pache JC, Soccal PM, Kaiser L. A prospective hospital-based study of the clinical impact of non-severe acute respiratory syndrome (Non-SARS)-related human coronavirus infection. Clin Infect Dis. 2006 Oct 15;43(8):1009-15. doi: 10.1086/507898. Epub 2006 Sep 13. PMID 16983613
- [Background] Cordero E, Aydillo T, Farinas MC, Pano-Pardo JR, Pachon J, Viasus D, Riera M, Lopez-Medrano F, Payeras A, Moreno A, Rodriguez-Bano J, Oteo JA, Martinez-Montauti J, Torre-Cisneros J, Segura F, Carratala J; Novel Influenza A(H1N1) Study Group of the SpanishNetwork for Research in Infectious Diseases (REIPI). Immunosuppressed patients with pandemic influenza A 2009 (H1N1) virus infection. Eur J Clin Microbiol Infect Dis. 2012 Apr;31(4):547-56. doi: 10.1007/s10096-011-1346-3. Epub 2011 Jul 27. PMID 21792558
- [Background] Tian S, Hu N, Lou J, Chen K, Kang X, Xiang Z, Chen H, Wang D, Liu N, Liu D, Chen G, Zhang Y, Li D, Li J, Lian H, Niu S, Zhang L, Zhang J. Characteristics of COVID-19 infection in Beijing. J Infect. 2020 Apr;80(4):401-406. doi: 10.1016/j.jinf.2020.02.018. Epub 2020 Feb 27. PMID 32112886
- [Background] Teicher E, Vincent I, Bonhomme-Faivre L, Abbara C, Barrail A, Boissonnas A, Duclos-Vallee JC, Taburet AM, Samuel D, Vittecoq D. Effect of highly active antiretroviral therapy on tacrolimus pharmacokinetics in hepatitis C virus and HIV co-infected liver transplant recipients in the ANRS HC-08 study. Clin Pharmacokinet. 2007;46(11):941-52. doi: 10.2165/00003088-200746110-00002. PMID 17922559
- [Background] Jain AB, Venkataramanan R, Eghtesad B, Marcos A, Ragni M, Shapiro R, Rafail AB, Fung JJ. Effect of coadministered lopinavir and ritonavir (Kaletra) on tacrolimus blood concentration in liver transplantation patients. Liver Transpl. 2003 Sep;9(9):954-60. doi: 10.1053/jlts.2003.50171. PMID 12942457
- [Background] Sheikh AM, Wolf DC, Lebovics E, Goldberg R, Horowitz HW. Concomitant human immunodeficiency virus protease inhibitor therapy markedly reduces tacrolimus metabolism and increases blood levels. Transplantation. 1999 Jul 27;68(2):307-9. doi: 10.1097/00007890-199907270-00027. PMID 10440408